CLINICAL TRIAL: NCT03412578
Title: Effect of Tactile/Kinaesthetic Massage Therapy on Growth Parameters and Body Composition of Preterm Infants
Brief Title: Effect of Tactile/Kinaesthetic Massage Therapy on DXA Parameter of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Associate Professor, Mansoura University Children Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NICU MUCH 2017
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Preterm Infant; Body Composition; Dual X-ray Absorptiometry (DXA) Scan
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Infants in this group will receive ordinary supportive care and will not receive Massage Therapy
- Massage group (Active Comparator): Infants in this group will receive Massage Therapy Massage therapy was started at corrected gestational age of 35 weeks and continued for 5 consecutive days. The protocol of massage therapy was performed as been described by Tiffany Field (Field, Schanberg et al. 1986). Three consecutive, 15 minutes, sessions were performed daily after the noon feeding. Each treatment session was divided into 5 minutes of tactile stimulation, followed by 5 minutes of kinaesthetic stimulation, and then another 5 minutes of tactile stimulation (Field, Diego et al. 2006).
  During massage therapy, infant's behavioural reaction was observed for signs of distress (e.g., yawning, finger splaying, crying).
  Interventions: Procedure: Massage Therapy

INTERVENTIONS:
Procedure: Massage Therapy — Massage therapy was started at corrected gestational age of 35 weeks and continued for 5 consecutive days. The protocol of massage therapy was performed as been described by Tiffany Field (Field, Schanberg et al. 1986). Three consecutive, 15 minutes, sessions were performed daily after the noon feeding. Each treatment session was divided into 5 minutes of tactile stimulation, followed by 5 minutes of kinaesthetic stimulation, and then another 5 minutes of tactile stimulation (Field, Diego et al. 2006).
  Arms: Massage group

SUMMARY:
The effect of Tactile/Kinaesthetic massage therapy on weight gain and different components of growth, as assessed by anthropometric measurements and DXA scan, and correlate these components with serum IGF-1, leptin and adiponectin in preterm infants.

DETAILED DESCRIPTION:
Prospective open label randomized, single-blind, controlled trial was done in the NICU at Mansoura University Children's Hospital.

Stable preterm infants in the NICU awaiting for sustained pattern of weight gain were included in the study.

Massage therapy was started at corrected gestational age of 35 weeks and continued for 5 consecutive days. The protocol of massage therapy was performed as been described by Tiffany Field. Three consecutive, 15 minutes, sessions were performed daily after the noon feeding. Each treatment session was divided into 5 minutes of tactile stimulation, followed by 5 minutes of kinaesthetic stimulation, and then another 5 minutes of tactile stimulation.

During massage therapy, infant's behavioural reaction was observed for signs of distress (e.g., yawning, finger splaying, crying). Vital signs are measured 15 minutes before, 15 minutes during and 15 minutes after the massage procedure. If signs of physiologic distress developed (heart rate greater than 200 bpm), massage was discontinued for 15 seconds, or until a return to baseline levels.

The study was discontinued if five periods of observed behavioural or physiological stress occurred.

Body composition assessment using DXA scan was performed for total body All infants were studied on one occasion by the end of 5 days massage therapy. DXA scan was performed without sedation but a pacifier with non-metallic parts was used as needed. The scanning procedure was interrupted if movement artefacts is noted. In addition, analyses of different body regions were also performed. Regional analyses typically involved the head, each of the four extremities, and the trunk.

Blood samples were collected using standard technique at baseline and after 5 days for measurement of IGF-1, leptin and adiponectin levels using Enzyme-linked Immunosorbent Assay [ELISA kit supplied by Elabscience Biotechnology (No.1 Shizishan Street, Wuhan, Hubei, China) catalog No: E-EL-H0086].

Randomization Infants were assigned randomly, by a designated neonatologist, to treatment groups using internet based random table technique with cards in opaque sealed envelopes that were kept in the neonatal care unit. A written informed consent was obtained from the parents of each infant upon enrolment in the study. Procedures of MT, DXA scan, and laboratory analysis were performed by a designated personnel throughout the study to ensure consistency. Performers of DXA scan and laboratory measures were blinded to groups of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable premature infants with gestational age at 28 to 37 weeks' admitted to the "grower" (step-down) nursery. Stability is defined as lack of need for supplemental oxygen, apneas and bradycardias, systemic antimicrobial therapy for infection, or a central line. On at least 100 ml/kg/d of feed (oral or tube feed) preterm formula. informed consent will be obtained from parents before enrollment in the study.

Exclusion Criteria:

* History of necrotizing enterocolitis, receipt of postnatal steroids, active infection, congenital malformations, chromosomal abnormality, intracranial hemorrhage more than (>) grade 2, inborn errors of metabolism, meningitis or encephalopathy, need for surgery.

Ages: 35 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Growth parameter (Weight) | 5 days
  Daily weight gain in grams and cumulative weight gain after 5 days of intervention
Growth parameter (Length) | 5 days
  Daily length gain in cm and cumulative length gain after 5 days of intervention
Growth parameter (Head circumference) | 5 days
  Daily head circumference gain in cm and cumulative head circumference gain after 5 days of intervention
Growth parameter (Mid-arm circumference) | 5 days
  Daily mid-arm circumference gain in cm and cumulative mid-arm circumference gain after 5 days of intervention
Growth parameter (Ponderal Index) | 5 days
  Daily changes in Ponderal Index and cumulative changes in Ponderal Index after 5 days of intervention

SECONDARY OUTCOMES:
Dual X-ray absorptiometry scan (DXA scan) | 5 days
  DXA scan will be performed prior to and 5 days after massage therapy to measure bone mineral density at different levels in the body
Insulin-like Growth Factor 1 (IGF-1) | 5 days
  Serum level of IGF-1 will be measured at baseline and 5 days after massage therapy
Serum Leptin | 5 days
  Serum level of Leptin will be measured at baseline and 5 days after massage therapy
Serum adiponectin | 5 days
  Serum level of adiponectin will be measured at baseline and 5 days after massage therapy

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura university children hospital, Al Mansurah, El Dakahlya
  - Al Mansurah

IPD SHARING:
Plan to Share IPD: Undecided